CLINICAL TRIAL: NCT01334242
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Determine the Pharmacodynamics of LX4211 Relative to Meals in Healthy Subjects
Brief Title: A Study to Determine the Pharmacodynamics of LX4211 Relative to Meals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Ikenna Ogbaa, MD - Medical Director, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-104-NRM; LX4211.104 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-04-06; First posted 2011-04-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LX4211 (Experimental): 400 mg of LX4211 administered orally
  Interventions: Drug: Schedule A; Drug: Schedule B; Drug: Schedule C; Drug: Schedule D; Drug: Schedule E
- Placebo (Placebo Comparator): Nonidentical placebo administered orally
  Interventions: Drug: Schedule A; Drug: Schedule B; Drug: Schedule C; Drug: Schedule D; Drug: Schedule E

INTERVENTIONS:
Drug: Schedule A — Dosing 1 hour before breakfast
Drug: Schedule B — Dosing 0.5 hour before breakfast
Drug: Schedule C — Dosing immediately before breakfast
Drug: Schedule D — Dosing immediately before lunch
Drug: Schedule E — Split dose, dosing 1 hour before breakfast and dinner

SUMMARY:
The primary purpose of this study is to evaluate the pharmacodynamics of LX4211 relative to meals in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 and ≤55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mm Hg; diastolic blood pressure, 50-90 mm Hg; heart rate, 50-100 bpm
* Body mass index (BMI) ≥18 and ≤35 kg/sq m
* Able to provide written informed consent

Exclusion Criteria:

* Use of any medication (prescription, over-the-counter, herbal tea, or supplements) within 5 days of dosing
* Use of any investigational agent or study treatment within 30 days of Day 1
* Use of any protein or antibody-based therapeutic agents within 3 months of Screening
* Prior exposure to any SGLT inhibitor
* Use of cigarettes or any tobacco products within 6 weeks prior to Screening and while participating in the study
* History of bariatric surgery or any other gastrointestinal surgery that may induce malabsorption
* History of any major surgery within 6 months of Screening
* History of any hypersensitivity to the inactive components of LX4211
* History of renal disease or significantly abnormal kidney function tests
* History of hepatic disease or significantly abnormal liver function tests
* History of any active infection within 30 days of Day 1
* History of alcohol or substance abuse within 2 years prior to Day 1
* Positive urine glucose at Screening
* Positive pregnancy test at Screening
* Inability or difficulty swallowing whole tablets or capsules
* Unable or unwilling to communicate or cooperate with the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Urinary glucose excretion | 24 hours collection on Day -1 and Days 7-13
Fasting Plasma Glucose | Day -1 and Days 7-12
Postprandial Glucose | Day -1 and Days 7-12
Insulin | Day -1 and Days 7-12
Glucagon-like peptide 1 (total and active) | Day -1 and Days 7-12
Peptide YY | Day -1 and Days 7-12

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Day 1 to Day 14
Blood chemistry | Day -2, Day 7 and Day 13
  Including albumin, ALP, ALT, AST, total bilirubin, glucose, BUN, calcium, carbon dioxide, chloride, cholesterol and triglycerides, creatinine, magnesium, phosphorus, potassium, sodium, protein, and uric acid.
Hematology | Day -2, Day 7 and Day 13
  Including complete blood count with differential, hemoglobin, hematocrit, lymphocyte, and platelet counts.

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zambrowicz B, Ogbaa I, Frazier K, Banks P, Turnage A, Freiman J, Boehm KA, Ruff D, Powell D, Sands A. Effects of LX4211, a dual sodium-dependent glucose cotransporters 1 and 2 inhibitor, on postprandial glucose, insulin, glucagon-like peptide 1, and peptide tyrosine tyrosine in a dose-timing study in healthy subjects. Clin Ther. 2013 Aug;35(8):1162-1173.e8. doi: 10.1016/j.clinthera.2013.06.011. Epub 2013 Jul 31. PMID 23911260